CLINICAL TRIAL: NCT04671615
Title: DEMOGRAPHICS, PATIENT CHARACTERISTICS, TREATMENT PATTERNS AND CLINICAL OUTCOMES OF PATIENTS TREATED WITH PALBOCICLIB IN A REAL LIFE SETTING IN ISRAEL
Brief Title: A Study to Understand the Treatment Patterns and Patients and Their Clinical Outcomes Who Are Taking Palbociclib in a Real Life Setting in Israel.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481160; NCT04671615 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2020-11-24; First posted 2020-12-17 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer
Keywords: hormone receptor; positive/human epidermal growth factor 2 - negative (HR+/HER2-)
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with metastatic, HR+/HER2- breast cancer.: Patients who initiated first or subsequent lines of treatment with palbociclib
  Interventions: Drug: palbociclib

INTERVENTIONS:
Drug: palbociclib — As provided in real world practice
  Other Names: Ibrance

SUMMARY:
The purpose of this study is to understand the treatment patterns, patients and their clinical outcomes in a real life setting in Israel. This study was done in adult breast cancer patients who have started palbociclib combination treatment as per the national basket of health services in January 2018 until August 2020 for all lines of therapy.

This study had included adult patients who were prescribed with palbociclib for their breast cancer which had spread to other parts of the body.

Patients are followed for around 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of metastatic breast cancer, based on the National/MHS cancer registry.
* Newly diagnosed metastatic breast cancer patients and newly treated with palbociclib within 6 months of diagnosis, in any line of treatment in the metastatic setting.
* Available data on palbociclib treatment for at least 6 months.
* Continuous healthcare plan enrolment in MHS for at least one year before index date.

Exclusion Criteria:

* Patients that initiated HER2 inhibitors.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a population based retrospective database study that will include patients with metastatic, HR+/ HER2- breast cancer and who initiated first or subsequent lines of treatment with palbociclib. Data will be available from Maccabi Healthcare Services (MHS) database in Israel for patients who received approval for treatment with palbociclib since 01 January 2018 until 31 August 2020.
Sampling Method: Non-Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Pharmaceuticals Israel Ltd., Herzliya Pituah, Israel

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Moser SS, Mazursky OF, Shalev H, Apter L, Chodick G, Siegelmann-Danieli N. Real-world outcomes of patients with metastatic endocrine-responsive breast cancer receiving palbociclib-based combinations. Future Oncol. 2023 Jul;19(21):1473-1483. doi: 10.2217/fon-2023-0176. Epub 2023 Aug 2. PMID 37529919
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective data from Israel participants with hormone receptor positive (HR+)/ human epidermal growth factor receptor 2 negative (HER2-) metastatic breast cancer and who initiated first or subsequent lines of palbociclib along with combination treatment (aromatase inhibitor [AI] or fulvestrant) and had at least 24 months of follow up post treatment initiation were planned to be observed.
Pre-assignment Details: Data were identified and retrieved from Maccabi healthcare services (MHS) database for eligible participants who initiated palbociclib combination treatment from 01 January 2018 to 30 June 2020. The observation period was extended up to 30 June 2022 to include the follow up duration of minimum of 24 months post treatment initiation. Data was observed and evaluated during 18 months of this retrospective study (06 December 2020 to 30 June 2022) of this study.
Groups:
- Palbociclib: Participants with HR+/HER2- metastatic breast cancer, who had initiated palbociclib combination treatment in real world clinical practice as per the national basket of health services, were observed during this population based retrospective database study.
Period: Overall Study
Arm/Group | Palbociclib
Started | 559
Completed | 559
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants whose data were included and observed in the study.
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 65.00 [54.00 to 72.00]
Age, Customized [Count of Participants; unit: Participants]
  <=65 Years | 278
  >65 Years | 281
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 554
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: Kilogram per meter square] | 27.85 [24.65 to 31.83]
Number of Participants Categorized According to BMI [Count of Participants; unit: Participants] — Number of participants were classified according to BMI as underweight (BMI less than [<]18.50 kilogram per meter square [kg/m^2]), normal (BMI 18.50-24.99 kg/m^2), overweight (BMI 25.00-29.99 kg/m^2), obese (BMI greater than or equal to [>=] 30 kg/m^2) and missing.
  Participants
    Underweight | 9
    Normal | 138
    Overweight | 190
    Obese | 186
    Missing | 36
Number of Participants According to Smoking History [Count of Participants; unit: Participants] — Number of participants were classified according to smoking history as current or former and never
  Participants
    Current or former | 210
    Never | 349
Number of Participants According to Region of Residence [Count of Participants; unit: Participants] — Number of participants according to region of residence included north, south and central region were reported.
  Participants
    North | 99
    South | 81
    Central | 379
Number of Participants According to Socioeconomic Status [Count of Participants; unit: Participants] — Number of participants were classified according to socioeconomic status as low, medium and high.
  Participants
    Low | 212
    Medium | 108
    High | 239
Number of Participants With Co-morbidities Diagnosed in one Year Prior to Palbociclib Initiation [Count of Participants; unit: Participants] — Participants with their co-morbidities diagnosed 1 year prior to palbociclib initiation were reported. One participant could have more than 1 co-morbidity so 1 participant could be included in more than 1 row reported below.
  Participants
    Diabetes mellitus | 133
    Cardiovascular disease | 76
    Ischemic heart disease | 27
    Hypertension | 279
    Chronic obstructive pulmonary disease (COPD) | 33
    Osteoporosis | 165
    Menopause | 439
Number of Participants With Chronic Disease - Depression [Count of Participants; unit: Participants] — Number of participants with depression as defined by international classification of diseases, ninth revision (ICD-9) codes were reported below.
  Participants | 174
Number of Participants According to Deyo-Charlson Comorbidity Index Categories [Count of Participants; unit: Participants] — Deyo-Charlson co-morbidity index was used to determine presence/absence of disease using international classification of diseases, ninth revision, clinical modification (ICD-9-CM) codes and MHS registries. It was calculated based on the presence of 19 comorbidities which have been selected and weighted on the basis of the strength of their association with mortality. Total score ranged from 0 to 9. A score of zero indicated that no comorbidities were found. The higher the score, the more likely the cumulative severity of a participant's comorbidities.
  Participants
    0 | 241
    1-2 | 205
    >=3 | 113
Number of Participants who Used Other Medications Prior to Palbociclib Initiation [Count of Participants; unit: Participants] — Number of participants who used other medications i.e. other than palbociclib (at least 2 purchases) within 3 months prior to index date (palbociclib initiation) were included.
  Participants | 0
Number of Participants who Visited Community/Hospital for Genetic Counselling [Count of Participants; unit: Participants] — Number of participants who visited community/hospital for genetic counselling for germline breast cancer gene mutation (gBRCAm) before index date were reported. Index date is date for initiation of palbociclib.
  Participants | 170
Number of Participants With Germline Breast Cancer Gene Mutation (gBRCAm) Test Performed [Count of Participants; unit: Participants] — Number of participants whose gBRCAm test was performed were reported.
  Participants | 164
Number of Participants According to Histology of Breast Cancer [Count of Participants; unit: Participants] — Number of participants according to histology of breast cancer as invasive ductal, invasive lobular, lobular and ductal and other/missing/unknown were reported.
  Participants
    Invasive ductal | 434
    Invasive lobular | 67
    Lobular and ductal | 19
    Other/missing/unknown | 39
Number of Participants According to Location of Metastases [Count of Participants; unit: Participants] — Number of participants according to location of metastases included visceral (lung, liver, abdomen or skin), lymph, bone and brain were reported. One participant could have more than 1 location so 1 participant could be included in more than 1 row.
  Participants
    Visceral | 261
    Lymph | 251
    Bone | 394
    Brain | 15
Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status was used to assess the physical health of participants and ranged from 0 to 5. where Grade 0: fully active; Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; Grade 2: ambulatory and capable of all self-care but unable to carry out any work activities; Grade 3: capable of only limited self-care; Grade 4: completely disabled. cannot carry on any selfcare and Grade 5: dead. Number of participants according to ECOG status were reported.
  Participants
    ECOG: 0-1 | 311
    ECOG: 2-4 | 70
    ECOG: Missing | 178
Number of Participants Categorized According to Hormone Receptor Sensitivity [Count of Participants; unit: Participants] — Number of participants according to hormone receptor sensitivity status included estrogen receptor positive (ER+)/ progesterone receptor positive (PR+), ER+, PR+ and missing were reported.
  Participants
    ER+/PR+ | 405
    ER+ | 139
    PR+ | 4
    Missing | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized According to Type of Index Combination Treatment Regimen
Description: Number of participants were classified on the basis of type of combination treatment along with palbociclib as first line therapy. Index treatment was palbociclib combination treatment. Index period was defined as duration in which participant initiated palbociclib combination treatment.
Time Frame: Day 1 of index treatment (any day from 01 January 2018 to 30 June 2020 [index period]), data observed and evaluated during 18 months of this retrospective study
Population: Analysis population included all participants whose data were included and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Participants
  Palbociclib + Aromatase Inhibitor (AI) | 293
  Palbociclib + Fulvestrant | 266

2. Primary Outcome: Duration of Index Treatment Per Type of Combination Treatment
Description: Duration in months between the start and stop of therapy was reported. Index treatment was palbociclib combination treatment. Kaplan-Meier method was used for the assessment of this outcome measure.
Time Frame: Day 1 of index treatment till discontinuation of index treatment (during 01 January 2018 to 30 June 2022 [approximately 54 months]); data observed and evaluated during 18 months of this retrospective study
Population: Analysis population included all participants whose data were included and observed in the study. Here "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Months
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 30.5 [23.7 to 37.2]
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant | 12.6 [10.6 to 15.6]

3. Primary Outcome: Number of Participants Categorized According to Number of Cycles of Index Treatment Per Type of Combination Treatment
Description: Number of participants categorized according to number of cycles of treatment including less than or equal to (<=) 6, greater than (>) 6 to 11, >11 to 20 and >20 cycles were reported. Index treatment was palbociclib combination treatment.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI: <= 6 cycles | 44
  Palbociclib + AI: >6 - 11 cycles | 37
  Palbociclib + AI: >11 - 20 cycles | 66
  Palbociclib + AI: >20 cycles | 146
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant: <= 6 cycles | 99
  Palbociclib + Fulvestrant: >6 - 11 cycles | 47
  Palbociclib + Fulvestrant: >11 - 20 cycles | 52
  Palbociclib + Fulvestrant: >20 cycles | 68

4. Primary Outcome: Number of Participants Categorized According to Initial Palbociclib Dose Per Type of Combination Treatment
Description: Number of participants were categorized according to initial palbociclib dose. Index treatment was palbociclib combination treatment. Index period was defined as duration in which participant initiated palbociclib combination treatment.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI: 75 milligrams (mg) | 8
  Palbociclib + AI: 100 mg | 23
  Palbociclib + AI: 125 mg | 262
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant: 75 milligrams (mg) | 12
  Palbociclib + Fulvestrant: 100 mg | 26
  Palbociclib + Fulvestrant: 125 mg | 228

5. Primary Outcome: Number of Participants With Modification (Reduction) in Initial Palbociclib Dose Per Type of Combination Treatment
Description: Number of participants who had a reduction in initial palbociclib dose were reported. Index treatment was palbociclib combination treatment.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 96
  Palbociclib+ Fulvestrant: number analyzed (Participants) | 266
  Palbociclib+ Fulvestrant | 82

6. Primary Outcome: Time on Treatment for Subsequent Treatment After Palbociclib Therapy Per Type of Combination Treatment
Description: Subsequent treatment after palbociclib therapy was the regimen received by participants following discontinuation from the palbociclib treatment and included chemotherapy, everolimus, fulvestrant and other. The duration between the start and stop of the post-palbociclib treatment was reported in this outcome measure. Index treatment was palbociclib combination treatment. Kaplan-Meier method was used for the assessment of this outcome measure.
Time Frame: Day 1 of subsequent treatment till last dose of subsequent treatment (during 01 January 2018 to 30 June 2022 [approximately 54 months]); data observed and evaluated during 18 months of this retrospective study
Population: Analysis population included all participants whose data were included and observed in the study. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure. All participants reported under "Overall Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 324
Months
  Palbociclib + AI: Chemotherapy: number analyzed (Participants) | 49
  Palbociclib + AI: Chemotherapy | 5.19 [3.16 to 8.55]
  Palbociclib + AI: Everolimus: number analyzed (Participants) | 30
  Palbociclib + AI: Everolimus | 4.57 [2.6 to 7.07]
  Palbociclib + AI: Fulvestrant: number analyzed (Participants) | 52
  Palbociclib + AI: Fulvestrant | 4.41 [3.72 to 6.08]
  Palbociclib + AI: Other: number analyzed (Participants) | 13
  Palbociclib + AI: Other | 12.89 [3.45 to NA] — Upper limit of 95% CI has not been reached due to less number of participants with events.
  Palbociclib + Fulvestrant: Chemotherapy: number analyzed (Participants) | 100
  Palbociclib + Fulvestrant: Chemotherapy | 6.08 [4.24 to 8.32]
  Palbociclib + Fulvestrant: Everolimus: number analyzed (Participants) | 58
  Palbociclib + Fulvestrant: Everolimus | 4.44 [3.06 to 6.38]
  Palbociclib + Fulvestrant: Fulvestrant: number analyzed (Participants) | 19
  Palbociclib + Fulvestrant: Fulvestrant | 7.76 [3.02 to NA] — Upper limit of 95% CI has not been reached due to less number of participants with events.
  Palbociclib + Fulvestrant: other: number analyzed (Participants) | 3
  Palbociclib + Fulvestrant: other | 4.37 [1.74 to NA] — Upper limit of 95% CI has not been reached due to less number of participants with events.

7. Primary Outcome: Percentage of Participants With Ongoing Index Treatment at Month 6 Per Type of Combination Treatment
Description: Percentage of participants with ongoing index treatment at Month 6 were reported. Index treatment was palbociclib combination treatment.
Time Frame: Day 1 of index treatment up to Month 6 of index treatment (during 01 January 2018 to 30 June 2022 [approximately 54 months]); data observed and evaluated during 18 months of this retrospective study
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Percentage of Participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 91.0 [87.7 to 94.3]
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant | 71.1 [65.7 to 76.9]

8. Primary Outcome: Percentage of Participants With Ongoing Index Treatment at Month 12 Per Type of Combination Treatment
Description: Percentage of participants with ongoing index treatment at Month 12 were reported. Index treatment was palbociclib combination treatment.
Time Frame: Day 1 of index treatment up to Month 12 of index treatment (during 01 January 2018 to 30 June 2022 [approximately 54 months]); data observed and evaluated during 18 months of this retrospective study
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Percentage of Participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 76.3 [71.5 to 81.4]
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant | 51.2 [45.2 to 57.9]

9. Primary Outcome: Percentage of Participants With Ongoing Index Treatment at Month 24 Per Type of Combination Treatment
Description: Percentage of participants with ongoing index treatment at Month 24 were reported. Index treatment was palbociclib combination treatment.
Time Frame: Day 1 of index treatment up to Month 24 of index treatment (during 01 January 2018 to 30 June 2022 [approximately 54 months]); data observed and evaluated during 18 months of this retrospective study
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Percentage of participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 54.7 [49.1 to 60.9]
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant | 26.0 [20.8 to 32.5]

10. Primary Outcome: Number of Participants Who Died Following Initiation of Index Treatment up to Month 6 Per Type of Combination Treatment
Description: Number of participants who died following index treatment up to Month 6 were reported. Index treatment was palbociclib combination treatment.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 10
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant | 31

11. Primary Outcome: Number of Participants Who Died Following Initiation of Index Treatment up to Month 12 Per Type of Combination Treatment
Description: Number of participants who died following index treatment up to Month 12 were reported. Index treatment was palbociclib combination treatment.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 21
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant | 71

12. Primary Outcome: Number of Participants Who Died Following Initiation of Index Treatment up to Month 24 Per Type of Combination Treatment
Description: Number of participants who died following index treatment up to Month 24 were reported. Index treatment is palbociclib combination treatment.
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Participants
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 58
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant | 119

13. Primary Outcome: Number of Participants Who Advanced and Did Not Advance to a Subsequent Treatment up to Month 6 Per Type of Combination Treatment
Description: Subsequent treatment after palbociclib therapy was the regimen received by participants following discontinuation from the palbociclib treatment. Number of participants who advanced and did not advance to a subsequent treatment up to Month 6 were reported. Index treatment is palbociclib combination treatment.
Time Frame: as for outcome 7
Population: Analysis population included all participants whose data were included and observed in the study. Here "Overall Number of Participants Analyzed" signifies participants evaluable for the outcome measure. All participants reported under "Overall Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 466
Participants
  Palbociclib + AI: number analyzed (Participants) | 224
  Palbociclib + AI: Advanced | 207
  Palbociclib + AI: Did not advance | 17
  Palbociclib + Fulvestrant: number analyzed (Participants) | 242
  Palbociclib + Fulvestrant: Advanced | 230
  Palbociclib + Fulvestrant: Did not advance | 12

14. Primary Outcome: Number of Participants Who Advanced and Did Not Advance to a Subsequent Treatment up to Month 12 Per Type of Combination Treatment
Description: Subsequent treatment after palbociclib therapy was the regimen received by participants following discontinuation from the palbociclib treatment. Number of participants who advanced and did not advance to a subsequent treatment up to Month 12 were reported. Index treatment is palbociclib combination treatment.
Time Frame: as for outcome 8
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 466
Participants
  Palbociclib + AI: number analyzed (Participants) | 224
  Palbociclib + AI: Advanced | 219
  Palbociclib + AI: Did not advance | 5
  Palbociclib + Fulvestrant: number analyzed (Participants) | 242
  Palbociclib + Fulvestrant: Advanced | 239
  Palbociclib + Fulvestrant: Did not advance | 3

15. Primary Outcome: Number of Participants Who Advanced and Did Not Advance to a Subsequent Treatment up to Month 24 Per Type of Combination Treatment
Description: Subsequent treatment after palbociclib therapy was the regimen received by participants following discontinuation from the palbociclib treatment. Number of participants who advanced and did not advance to a subsequent treatment up to Month 24 were reported. Index treatment is palbociclib combination treatment.
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 466
Participants
  Palbociclib + AI: number analyzed (Participants) | 224
  Palbociclib + AI: Advanced | 223
  Palbociclib + AI: Did not advance | 1
  Palbociclib + Fulvestrant: number analyzed (Participants) | 242
  Palbociclib + Fulvestrant: Advanced | 242
  Palbociclib + Fulvestrant: Did not advance | 0

16. Primary Outcome: Time to Initiation of Chemotherapy After Cessation of Initial Palbociclib Therapy Per Type of Combination Treatment
Description: Time to initiation of chemotherapy was the duration from end of index treatment up to start of chemotherapy. Index treatment is palbociclib combination treatment.
Time Frame: From cessation of index treatment up to initiation of chemotherapy (during 01 January 2018 to 31 December 2020 [approximately 36 months]); data observed and evaluated during 18 months of this retrospective study
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 116
Months
  Palbociclib + AI: number analyzed (Participants) | 32
  Palbociclib + AI | 0.79 [0.59 to 1.51]
  Palbociclib + Fulvestrant: number analyzed (Participants) | 84
  Palbociclib + Fulvestrant | 0.92 [0.79 to 1.118]

17. Primary Outcome: Time to Initiation of Next Treatment (TTNT) From Initiation of Palbociclib Treatment Per Type of Combination Treatment
Description: TTNT was defined as the interval between the start of the index treatment date and the date of the next-line treatment. Participants who did not advance to the next treatment were censored on the study end date or death, whichever occurred first. Index treatment is palbociclib combination treatment. Kaplan-Meier method was used for the assessment of this outcome measure.
Time Frame: Day 1 of index treatment up to initiation of next treatment (during 01 January 2018 to 30 June 2022 [approximately 54 months]); data observed and evaluated during 18 months of this retrospective study
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 559
Months
  Palbociclib + AI: number analyzed (Participants) | 293
  Palbociclib + AI | 34.5 [27.2 to 51.6]
  Palbociclib + Fulvestrant: number analyzed (Participants) | 266
  Palbociclib + Fulvestrant | 16.4 [13.3 to 18.1]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Any death due to any cause that happened was recorded during observation period from 01 January 2018 to 30 June 2022 (approximately 54 months); data observed and evaluated during 18 months of this retrospective study. Due to non-interventional nature of the study adverse events were not collected and recorded, hence time frame not applicable.
Description: Due to non-interventional nature of the study, data for SAEs and non-SAEs were not collected.
Arm/Group | Palbociclib
All-Cause Mortality (participants affected / at risk) | 269/559
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT04671615/Prot_SAP_001.pdf